CLINICAL TRIAL: NCT00646737
Title: Phase IV Study of Enteric-coated Mycophenolate Sodium in Combination With Tacrolimus in Renal Transplant Patient
Brief Title: Conversion From Mycophenolate Mofetil to Mycophenolate Sodium in Renal Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080ABR02
Record Dates: First submitted 2008-03-18; First posted 2008-03-28 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; conversion; mycophenolate mofetil; mycophenolate sodium,; tacrolimus
MeSH Terms: interventions — Mycophenolic Acid

ARMS (1):
- 1 (Experimental): Mycophenolate sodium
  Interventions: Drug: Mycophenolate sodium

INTERVENTIONS:
Drug: Mycophenolate sodium — Mycophenolate sodium

SUMMARY:
The purpose of this study is to evaluate the safety and the tolerability of the substitution of mycophenolate mofetil for enteric-coated mycophenolate sodium in a population of stable renal transplant patients in Brazil, in a treatment regimen of immunosuppressants with tacrolimus and mycophenolate mofetil.

ELIGIBILITY:
Inclusion criteria

* Age between 18 and 65 years;
* First or second renal transplant within at least 12 weeks;
* Clinical stability, in the opinion of the investigator, during at least 8 weeks before inclusion in the study;
* Women of reproductive age must use contraceptive methods and present negative results in pregnancy test Serum creatinine < 2.5 mg/dE; Patients in use of a immunosuppression regimen based on tacrolimus and mycophenolate mofetil (generic or not, in any dose), who present gastrointestinal symptoms Capacity to complete the study requirements;

Exclusion criteria History of acute rejection,

* Proven or not by biopsy, in the last 2 months before the study;
* Recipients of multiple organs;
* Participation in any clinical investigation in the last 6 months before the present study;
* Thrombocytopenia (platelets <75,00O/mm3), leucopenia (total leukocytes <4,000/mm3)and/or anemia (hemoglobin <9.0 gldL) before inclusion in the study;
* Clinically important disease, in the opinion of the investigator, including systemic infection, within 2 weeks before inclusion in the study;
* Presence of any neoplasia, current or past, except resected basal cell carcinoma;
* Any surgical or medical condition that could significantly alter the absorption, distribution, metabolism or excretion of medicines or that could put the patient in danger as a result of participation in the study;
* History of drug or alcohol abuse within previous 12 months of inclusion in the study, Current or prior use in the last 2 months of bile acid-adsorbing resins(cholestyramine and colestipol).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal symptoms in renal transplant patients treated with the immunosuppression regimen of tacrolimus and mycophenolate at baseline, 8 and 16 weeks | 8 and 16 weeks

SECONDARY OUTCOMES:
Impact of gastrointestinal symptoms on quality of life. Tolerability of mycophenolate sodium in combination with tacrolimus assessed by OSRS. Safety of mycophenolate sodium in combination with tacrolimus assessed by incidence of adverse events | 8 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigative Site, São Paulo, Brazil

REFERENCES:
- [Result] Pacheco e Silva Filho A, Manfro RC, Contieri FL, Mazzali M, Garcia VD, Carvalho Dde B, David S, Machado P, Rodrigues CA. Evaluation of tolerability of enteric-coated mycophenolate sodium versus mycophenolate mofetil in de novo renal transplantation. J Bras Nefrol. 2015 Jul-Sep;37(3):291-6. doi: 10.5935/0101-2800.20150048. English, Portuguese. PMID 26398638